CLINICAL TRIAL: NCT01502280
Title: Barrow 5-ALA Intraoperative Confocal Evaluation Trial
Brief Title: Fluorescence-guided Surgery for Low- and High-grade Gliomas
Acronym: BALANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#10BN132
Record Dates: First submitted 2011-12-22; First posted 2011-12-30 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2017-01

CONDITIONS: Glioma
Keywords: extent of resection; Glioma; 5-ALA; tumor fluorescence; confocal microscopy
MeSH Terms: conditions — Glioma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-ALA/Gliolan® /5-Aminolevulinic acid (Experimental): Within 3 hours prior to surgery, patient will orally ingest [or be given via Nasogastric (NG), Orogastric (OG), or Gastric tube (G-tube)] 5-ALA/Gliolan®/5-Aminolevulinic acid mixed with sterile water (20mg/kg)
  Interventions: Drug: 5-Aminolevulinic acid (ALA)
- Placebo - ascorbic acid (Placebo Comparator): Within 3 hours prior to surgery, patient will orally ingest [or be given via Nasogastric (NG), Orogastric (OG), or Gastric tube (G-tube)] 1.5 Gm. placebo - ascorbic acid in 50 ml sterile water.
  Interventions: Drug: Placebo - ascorbic acid

INTERVENTIONS:
Drug: 5-Aminolevulinic acid (ALA) — Following informed consent, within 3 hours prior to surgery, patient will orally ingest [or be given via Nasogastric (NG), Orogastric (OG), or Gastric tube (G-tube)] either (1) 5-ALA/Gliolan® mixed with sterile water (20mg/kg)
  Other Names: 5-Aminolevulinic acid Hydrochloride; Gliolan®; 5-ALA
  Arms: 5-ALA/Gliolan® /5-Aminolevulinic acid
Drug: Placebo - ascorbic acid — Within 3 hours prior to surgery, patient will orally ingest [or be given via Nasogastric (NG), Orogastric (OG), or Gastric tube (G-tube)] 1.5 Gm. placebo - ascorbic acid in 50 ml sterile water.
  Arms: Placebo - ascorbic acid

SUMMARY:
Gliomas are the most common primary brain tumor, yet remain a challenge to effectively treat. Mounting evidence suggests that survival improves with greater tumor removal, yet being able do a complete removal can be difficult due to the tumor's infiltrating nature. 5-aminolevulinic acid (5-ALA) is a natural compound that, when patients take it by mouth 3 hours before surgery, is selectively taken up by glioma cells and causes a red/pink fluorescence (glow) under a blue light that allows tumor margins to be seen during the course of surgery. While this compound is used as a standard-of-care agent in Europe, it remains under testing by the Food and Drug Administration (FDA). A recent clinical trial in Germany, however, has demonstrated a significant improvement in the rate of complete resection for certain brain tumors (65% vs. 34%).

The Barrow 5-ALA Intraoperative Confocal (BALANCE) Trial will measure the effect of 5-ALA on the amount of glioma tumor removal. To improve the usefulness of 5-ALA, a new special microscope fitted with a blue light, will be used to magnify microscopic fluorescence at the tumor margins. The investigators' hypothesis is that 5-ALA fluorescence with the use of the special microscope during surgery will greatly lower the amount of tumor left behind.

DETAILED DESCRIPTION:
Gliomas are the most common primary brain tumor, yet are associated with a 12-14 month overall survival in the United States. Mounting evidence suggests that survival improves with greater extent of resection, yet achieving a complete radiographic resection is challenging due to the tumor's infiltrating nature. Oral 5-aminolevulinic acid (5-ALA/Gliolan®) is a natural compound that, when administered to patients within 3 hours prior to surgery, is selectively metabolized by glioma cells and induces a red/pink fluorescence under blue light that facilitates intraoperative identification of tumor margins. While this compound is used as a standard-of-care agent in Europe, it remains under examination by the Food and Drug Administration (FDA). A recent multicenter randomized, single-blind, controlled study in Germany demonstrated a significant improvement in the rate of complete resection for high-grade gliomas, as compared to conventional microneurosurgery (65% vs. 34%) (Stummer et al., Lancet Oncology 2006).

Patients with presumed newly-diagnosed glioma will be entered into the trial. On the basis of their expected extent of resection (low vs. high), they will be stratified in one of 2 groups - Group 1 (expected high extent or resection) or Group 2 (expected low extent of resection). Following stratification, patients with newly-diagnosed disease will be randomized to receive either study drug (5-ALA/Gliolan®) or placebo (ascorbic acid) prior to surgery. Those who have had previous biopsy only without further treatment will be eligible for randomization. Intraoperatively, 5-ALA/Gliolan® patients will undergo resection with combined fluorescence microscopy and confocal microscopy. Placebo patients will undergo resection with standard light microscopy. Postoperatively, patients will have an MRI scan with and without contrast within 48 hours of surgery. Subsequent analysis of each patient will include assessment of the primary endpoint, that is,volume of residual disease (VRD) by volumetrically quantifying the tumor before and after surgery using T1-weighted contrast-enhancement (high-grade gliomas) or T2-weighted hyperintensity (low-grade gliomas). Similarly, volumetric extent of resection will also be measured. Other secondary endpoints will include overall survival (OS), progression-free survival (PFS), and National Institute of Health Stroke Scale (NIHSS) (collected at baseline, 7-10 days post-op and at 6, 12, 18, and 24 months post op).

The Barrow 5-ALA Intraoperative Confocal (BALANCE) study will quantify the impact of 5-ALA/Gliolan(R) on low- and high-grade glioma extent of resection. To enhance the efficacy of 5-ALA/Gliolan(R), particularly for low-grade gliomas that fluoresce less vigorously due to their comparatively lower cellular metabolism, intraoperative confocal microscopy will be used to amplify microscopic fluorescence at the tumor margins. The investigators' hypothesis is that, for both low- and high-grade gliomas, 5-ALA/Gliolan(R) fluorescence in conjunction with intraoperative confocal microscopy will significantly lower the VRD.

Goals:

1. To determine the impact of intraoperative fluorescence and confocal microscopy on the volume of residual disease following resection of a newly-diagnosed glioma.

Sub-goals:

1. To assess the feasibility and utility of combining intraoperative fluorescence with confocal microscopy.
2. To determine the impact of this combined approach in improving volumetric extent of resection.
3. To determine the impact of this combined approach in improving overall survival and 6-month progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Presumed newly-diagnosed supratentorial glioma (previous biopsy-only/no adjuvant therapy are eligible for randomization)
* Age > 18 years
* Normal bone marrow function (WBC > 3000, Platelets > 100,000)

Exclusion Criteria:

* Infratentorial tumors
* Pregnancy
* Hypersensitivity to 5-aminolevulinic acid hydrochloride or porphyrins
* History of photosensitivity, porphyria, or exfoliative dermatitis
* Hepatic dysfunction in the last 12 months (defined by AST, ALT, ALP, bilirubin > 2.5 x normal)
* Serum creatinine > 180 µmol/L
* Estimated Glomerular Filtration Rate (eGFR) < 60 ml/min/1.73m2
* Inability to undergo MRI scan with contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2010-11; Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Volumetric extent of resection | Change in MRI from pre-operative to within 48 hours post-operative
  Volumetric analysis of MRI contrast T1-weighted images (for low grade gliomas) will be compared to the preoperative sequences to calculate the volume of residual disease. Slice-by-slice assessment of pre- and postoperative tumor volume will be quantified by sequentially measuring the area of tumor on each slice and then integrating the combined measurements. This methodology has been previously reported (Sanai et al., Journal of Neurosurgery, 2010; Sanai et al, The New England Journal of Medicine, 2008)

SECONDARY OUTCOMES:
Overall Survival rate(OS) | Time from randomization until date of death assessed up to 48 months
  overall survival
Progression-free survival rate (PFS) | Time from randomization until first date of progression assessed up to 48 months
  time from surgery to progression
National Institute of Health Stroke Scale (NIHSS) | Change in score from pre-operative at post-operative, 6, 12, 18 and 24 months
  composite score

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — St. Joseph's Hospital Medical Center, Phoenix
Locations (1):
- St. Joseph's Hospital and Medical Center/Barrow Neurological Institute, Phoenix, Arizona, United States

REFERENCES:
- [Result] Sanai N, Snyder LA, Honea NJ, Coons SW, Eschbacher JM, Smith KA, Spetzler RF. Intraoperative confocal microscopy in the visualization of 5-aminolevulinic acid fluorescence in low-grade gliomas. J Neurosurg. 2011 Oct;115(4):740-8. doi: 10.3171/2011.6.JNS11252. Epub 2011 Jul 15. PMID 21761971